CLINICAL TRIAL: NCT05621759
Title: Phase II Single-Arm Open-Label Study Of Reduced-Dose Post-Transplant Cyclophosphamide, Abatacept, and Short-Duration Tacrolimus for the Prevention of Graft-Versus-Host Disease (GVHD) Following Haploidentical Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Cyclophosphamide, Abatacept, and Tacrolimus for the Prevention of GvHD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-00674
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Graft Vs Host Disease
Keywords: Haploidentical Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide; Abatacept; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Reduced-Dose Post-Transplant Cyclophosphamide, Abatacept, and Short-Duration Tacrolimus (Experimental): Participants to receive:
  * Cyclophosphamide 25 mg/kg IV over 1 hour on Day 3 and Day 4 following transplant
  * Abatacept 10 mg/kg IV on Day 5, Day 14, Day 28, and Day 56 following transplant
  * Tacrolimus 0.02 mg/kg IV by continuous infusion, starting on Day 5 following transplant. May switch to oral administration when tolerated, adjusted to maintain a drug level between 5-12ng/mL. Tacrolimus treatment is continued until Day 60 and then tapered over a period of 4 weeks in the absence of GvHD.
  Interventions: Drug: Cyclophosphamide; Drug: Abatacept; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Nitrogen mustard alkylating agent produced by Bristol-Myers Squibb.
  Other Names: Cytoxan
Drug: Abatacept — Calcineurin-inhibitor produced by Astellas.
  Other Names: Prograf
Drug: Tacrolimus — Selective T cell co-stimulation modulator produced by Bristol-Myers Squibb.
  Other Names: Orencia

SUMMARY:
This is a single arm, open label, phase II clinical trial. Adult patients with hematological malignancies undergoing allogeneic HSCT from first- or second-degree haploidentical donor are eligible for the study if they meet the standard criteria defined in our institutional standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Patients will receive non-myeloablative, reduced-intensity or myeloablative conditioning regimen followed by peripheral blood hematopoietic stem cells. Patients will receive dosed reduced cyclophosphamide, abatacept, and short-duration tacrolimus for GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky score ≥ 70%
* No evidence of progressive bacterial, viral, or fungal infection
* Creatinine clearance > 50 mL/min/1.72m2
* Total bilirubin, Alanine Aminotransferase and Aspartate Aminotransferase < 2 x the upper limit of normal (except for diagnosed Gilbert's syndrome)
* Alkaline phosphatase ≤ 250 IU/L
* Left Ventricular Ejection Fraction (LVEF) > 45%
* Adjusted Carbon Monoxide Diffusing Capacity (DLCO) > 60%
* Negative HIV serology
* Negative pregnancy test: confirmation per negative serum β-human chorionic gonadotropin (β-hCG) for women of childbearing age and potential.

Exclusion Criteria:

* Donors are excluded in case of donor-specific HLA antibodies or positive cross-match.
* Pregnant or nursing females or women of child bearing age or potential, who are unwilling to completely abstain from heterosexual sex or practice 2 effective methods of contraception from the first dose of conditioning regimen through day +180. A woman of reproductive capability is one who has not undergone a hysterectomy (removal of the womb), has not had both ovaries removed, or has not been post-menopausal (stopped menstrual periods) for more than 24 months in a row.
* Male subjects who refuse to practice effective barrier contraception during the entire study treatment period and through a minimum of 90 days after the last dose of study drug, or completely abstain from heterosexual intercourse. This must be done even if they are surgically sterilized (i.e., post-vasectomy).
* Inability to provide informed consent.
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix E), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Known allergies to any of the components of the investigational treatment regimen.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of Grades II-IV Acute GvHD | Up to Day 120
  The first day of acute GvHD of any grade is used to calculate the cumulative incidence for that grade. The diagnosis of acute GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.

SECONDARY OUTCOMES:
Cumulative Incidence of Chronic GvHD | Up to Day 365
  The first day of chronic GvHD is used to calculate the cumulative incidence of chronic GvHD. The diagnosis of chronic GvHD is based on clinical and pathological evaluation by the principal investigator in collaboration with the treating physician.
Number of Participants Presenting with Primary Graft Failure | Up to Day 45
  Primary graft failure is defined as failure to achieve neutrophil engraftment by Day 28 after transplant or lack of donor chimerism greater than 50% by Day 45, not due to the underlying malignancy.
Number of Participants Presenting with Poor Graft Function | Up to Day 30
  Poor graft function is defined by at least 2 of the following 3 criteria: Hemoglobin less than 8 g/dL, absolute neutrophil count less than 0.5 x 109/L, and platelets less than 20 x 109/L. The cytopenia must be unexplained (such as by disease relapse) and unresponsive to cytokines and must last at least 4 weeks.
Number of Participants Presenting with Secondary Graft Failure | Up to Day 730
  Secondary graft failure is defined as poor graft function associated with donor chimerism less than 5%.
Treatment-Related Mortality (TRM) Rate | Up to Day 730
  The proportion of participant deaths not attributable to disease relapse or progression.
Relapse Rate (RR) | Up to Day 730
  The proportion of participants in whom the disease for which transplant was performed is evident by methods of disease detection.
GvHD and Relapse-Free Survival (GRFS) Rate | Up to Day 730
  The proportion of participants who are without reported grade III-IV acute GvHD, chronic GvHD requiring systemic therapy and have not experienced relapse or death.
Overall Survival (OS) Rate | Up to Day 730
  The proportion of participants who are alive at the end of the study's evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Maher Abdul Hay, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only available to study team members.